CLINICAL TRIAL: NCT02130128
Title: Continuing Evaluation of the LungPoint ATV System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sufficient clinical evidence was gathered
Sponsor: Broncus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Protocol 42
Record Dates: First submitted 2014-04-28; First posted 2014-05-05 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Navigation and tissue sampling (Experimental): Guided bronchoscopic navigation and lung tissue sampling using the LungPoint ATV System
  Interventions: Device: LungPoint ATV System

INTERVENTIONS:
Device: LungPoint ATV System — The LungPoint ATV System is an image-guided navigation system used to access tissue samples in the lungs.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the LungPoint ATV System in patients who are scheduled for standard bronchoscopy to diagnose highly suspicious lung cancer.

DETAILED DESCRIPTION:
The LungPoint ATV System is an image-guided navigation system used to access tissue samples in the lungs. This feasibility study is being conducted to assess the safety and yield of the LungPoint ATV System in patients who are scheduled for standard bronchoscopy to diagnose highly suspicious lung cancer. Navigation to and sampling of the patient's lung cancer tumor is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical candidates age 21-75 years at screening
2. Highly suspicious SPN, defined as distinct nodule with a diameter of 10-30 mm in its largest dimension
3. No known endobronchial tumor
4. Tumor located anywhere in parenchymal tissue >1 cm from pleura and accessible bronchoscopically through a POE.
5. Willing to participate in all aspects of study protocol for duration of study
6. Able to understand study requirements
7. Signs study-related informed consent document

Exclusion Criteria:

1. Any contraindication to bronchoscopy, for example: (a.) Untreatable life-threatening arrhythmias, (b.) Inability to adequately oxygenate the patient during the procedure, (c.) Acute respiratory failure with hypercapnia (unless the patient is intubated and ventilated), (d.) Recent myocardial infarction, (e.) Previously diagnosed high-grade tracheal obstruction, (f.) Uncorrectable coagulopathy.
2. Known coagulopathy
3. Platelet dysfunction or platelet count < 100 x 103 cells/mm3
4. History of major bleeding with bronchoscopy
5. Pulmonary hypertension with mean PAP >25 mm
6. Moderate-to-severe pulmonary fibrosis
7. Moderate to severe emphysema or COPD with FEV1 <60% predicted or RV >200% predicted
8. Bullae >5 cm located in vicinity of target SPN or ATV tunnel
9. Any other severe or life-threatening comorbidity that could increase the risk of bronchoscopic biopsy or ATV tunneling, for example: (a.) ASA class > 3, (b.) > stage 3 heart failure, (c.) severe cachexia, (d.) severe respiratory insufficiency or hypoxia
10. Ongoing systemic infection
11. Contraindication to general anesthesia
12. Chronic use of anticoagulants (e.g., heparin, Warfarin) or antiplatelet agents (e.g. aspirin, clopidogrel)
13. Participation in any other study in last 30 days
14. Prior thoracic surgery on the same side of the lung as the SPN
15. Breastfeeding women or females of childbearing potential with a positive pregnancy test prior to the procedure or the intent to become pregnant during the study.
16. Life expectancy of less than one year.
17. Patients with known intrapulmonary metastases of extrapulmonary cancer/tumors
18. Scheduled for lung surgery within 7 days post-scheduled diagnostic bronchoscopy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse events | Up to 24 hours post procedure
  The number of serious adverse events (SAEs) rated as probably or definitely related to the study device and/or procedure divided by the number of patients in whom an attempt at study device use was made. This study protocol focuses specifically on sub-chronic pneumothorax, but will also track hemoptysis.

SECONDARY OUTCOMES:
Proportion of biopsies yielding tissue sufficient for diagnosis | Upon asssessment of histology of tissue sample taken during procedure
  The number of nodules with at least one biopsy sufficient for a tissue diagnosis divided by the number of nodules sampled by the LP ATV System.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, MD, Principal Investigator — Heidelberg University
Locations (1):
- Thoraxklinik, Heidelberg, Germany